CLINICAL TRIAL: NCT04212130
Title: The Effect of Fluorescent Marking and BCA Methods of Patient Unit Cleaning in Intensive Care
Brief Title: Can Environmental Cleanliness be Assessed by BCA (Bicinchoninic Acid) Method
Acronym: BCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zuhal Gülsoy, Lead researcher, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Cumhuriyet University
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Nosocomial Infection; Infection Control; Multi-antibiotic Resistance
Keywords: Intensive care unit; Infection Control; Microbiological Monitoring; High-touch surfaces; Fluorescent marker; Hospital environment; Cleanliness assessment
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of environmental cleanliness (Experimental): In this study,
  1. fluorescent marking,
  2. microbiological sampling and
  3. BCA methods will be compared in order to evaluate the effectiveness and usability of BCA method
  Interventions: Other: BCA method for assessing environmental cleanliness

INTERVENTIONS:
Other: BCA method for assessing environmental cleanliness — Evaluating the effectiveness and usability of BCA method which is a new approach in evaluating the effectiveness of environmental cleanliness in intensive care units.
  In this study, fluorecan labeling, microbiological sampling and BCA methods will be compared in order to evaluate the effectiveness and usability of BCA method
  Other Names: Pro 1 Micro Hygiene Monitoring Systems

SUMMARY:
Effective cleaning of surfaces in the hospital environment is an absolute necessity to reduce pathogen transmission. Multi Drug Resistant Organisms (MDRO) in ICU are among the leading causes of hospital-acquired infections. Today, the growing prevalence of MDRO has made it more important than ever to clean contaminated surfaces with appropriate aseptic cleaning procedures, to protect patients and personnel. Despite the disinfection and sterilization methods, microorganisms that reach a sufficient concentration in the hospital environment survive for long periods and can cause serious transmission via contaminated hands of healthcare workers. In this context, surface cleaning and disinfection procedures in the hospital environment reduce cross-contamination of the health care units and disease-causing pathogens. Recently, environmental cleaning and disinfection have become important as well as the evaluation of cleanliness.

The aim of this study is to evaluate the effectiveness and usability of BCA method, which is a new approach in evaluating the effectiveness of environmental cleanliness in intensive care units. fluoroscan gel marking, microbiological sampling and BCA assay methods will be compared to evaluate the effectiveness and usability of the BCA method. (PRO1 Micro Hygiene Monitoring System that System consisting of protein pen and device that analyzes with BCA method).

DETAILED DESCRIPTION:
Patients admitted to the ICU are at great risk of developing nosocomial infections, partly because of their serious illness and partly because of exposure to life-saving invasive procedures. In ICU, implementation of invasive procedures, with the purpose of diagnosis and treatment, such as urinary catheter, central-peripheral catheter, intubation, and being subject to intensive antibiotic use increase the likelihood of infection. Environmental cleanliness is important for preventing infections.

Effective cleaning of surfaces in the hospital environment is an absolute necessity to reduce pathogen transmission. Multi Drug Resistant Organisms (MDRO) in ICU are among the leading causes of hospital-acquired infections. Today, the growing prevalence of MDRO has made it more important than ever to clean contaminated surfaces with appropriate aseptic cleaning procedures, to protect patients and personnel. Despite the disinfection and sterilization methods, microorganisms that reach a sufficient concentration in the hospital environment survive for long periods and can cause serious transmission via contaminated hands of healthcare workers. In this context, surface cleaning and disinfection procedures in the hospital environment reduce cross-contamination of the health care units and disease-causing pathogens. Recently, environmental cleaning and disinfection have become important as well as the evaluation of cleanliness.

Cleaning of frequently contacted environmental surfaces, monitoring and verifying the cleaning results are important for patient safety. The effectiveness of environmental cleaning can be assay by different methods. Visual evaluation, ATP (AdenosineTriphosphate) measurement, protein tests and fluoroscan marking methods are some of them.

Evaluation of the patient unit cleanup in the ICU, that is carried out after the discharge of patients with infection or colonization that would require strict contact isolation, by Fluoroscan Marking, BCA and Microbiological Sampling methods, is planned with the aim of collecting data in order to prove the efficiency and clinical employability of the new cleaning assessment method, PRO1 Micro Hygiene Monitoring System (System consisting of protein pen and device that analyzes with BCA method).

ELIGIBILITY:
Inclusion Criteria:

A patient infected with resistant microorganism in the unit is in the same unit for at least 72 hours

The first BCA measurement when the unit is discharged gives a result indicating the unit is dirty.-

Exclusion Criteria:

* The patient who has been infected with the resistant microorganism in the unit has been hospitalized for less than 72 hours
* The first BCA measurement when the unit is empty does not give a result indicating that the unit is dirty.
* Impaired blindness for any reason included in the study
* In case the patient is included in the study but new patient admission to the unit before the cleaning stages are completed
* In the event that other employees who are included in the work but do not complete the cleaning stages enter and leave the unit, the work will be terminated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of cleaning | 1 year
  The absence of gel residue on the surfaces indicates that the wiping process is effective. Microbiological samples will determine the presence and amount of bacteria (colony) in the environment. It is aimed that bacteria cannot be produced in the samples taken from the environment after cleaning. The BCA protein samples will be analyzed by the researcher using the PRO 1 Micro hygiene monitoring device. PRO 1 Micro hygiene monitoring device will detect the presence of biological material on the surfaces. The presence and amount of bacteria on the surface will be determined with BCA protein. The presence and amount of bacteria can be detected by BCA protein swab, but not by bacterial species. The device is capable of detecting the biological load between 1 - 10 micrograms. Areas with values above 5 micrograms will be considered as dirty, areas with values below 5 micrograms will be considered as clean

SECONDARY OUTCOMES:
To evaluate the effectiveness of BCA method | 1 year
  If cleaning is not considered to be effective, cleaning will be repeated. If the results of samples taken with BCA protein pen after effective cleaning are below 5 microns, it is concluded that the area, is clean. If the BCA method (micrograms) shows clean or similar results in microbiological samples (colony), it will be concluded that the BCA method can be used to evaluate surface cleanliness.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)